CLINICAL TRIAL: NCT00863382
Title: Comparison of External Event Recorders With Implantable Monitor for Post Atrial Fibrillation Monitoring: Assessment of Cost and Efficacy
Brief Title: Comparison of External Event Recorders for Atrial Fibrillation Monitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Associate Professor of Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11566
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard Event Monitor
  Interventions: Device: Standard Event Monitor
- 2 (Active Comparator): Sleuth recorder
  Interventions: Device: Sleuth Monitor

INTERVENTIONS:
Device: Standard Event Monitor — Standard Event Monitor
  Arms: 1
Device: Sleuth Monitor — Implantable Sleuth Recorder
  Arms: 2

SUMMARY:
Ablation of atrial fibrillation is a well established treatment method to restore normal sinus rhythm and eliminate the need for continued antiarrhythmic therapy and anticoagulation. Absence of symptomatic and asymptomatic atrial fibrillation should be considered necessary for discontinuation of anticoagulation therapy. Presently, recurrence of atrial fibrillation is usually determined with the use of a non looping event monitor which is typically used by the subject at the time of symptomatic arrhythmia. This method does not detect asymptomatic atrial fibrillation. Random asymptomatic recording can be added, but the chance for detecting recurrence of arrhythmia is not great. Too frequently, the success rates of AF ablation procedures are inflated by insufficient follow up and patient's limited compliance in reporting and recording episodes of recurrent arrhythmias. Often times, it is very inconvenient for patients to wear external event recorders. Allergies to the sticky pads that are needed for most of the external monitoring devices continues to be a problem. Implantable loop recorders have the advantage of detecting symptomatic and asymptomatic atrial fibrillation continuously. They also offer the convenience of monitoring for up to 18 to 24 months without significant patient discomfort. However, implantation and explantation of these devices involves a limited surgical procedure as well as considerable experience. In this study we attempt to assess the differences in these two types of monitoring systems in assessing the long term efficacy of AF ablation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who undergo radiofrequency ablation of paroxysmal AF.

Exclusion Criteria:

* Subjects with known allergy to sticky patches of event monitor
* Subjects with skin infection or other problems on the chest that interferes with monitor implantation
* Subjects who are scheduled for radiation therapy
* Subjects who are scheduled for therapeutic ultrasound (like lithotripsy)
* Subjects who are scheduled for MRI
* Subjects who are scheduled for a procedure that uses diathermy.
* Subjects, in the opinion of the investigator, are not suitable candidates for the study
* Subjects that do not have analog telephone line at home.
* Existing Cardiac Rhythm Management Device (e.g., pacemaker or ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
recurrence of atrial fibrillation | 6 months, 1 year, 2 years

SECONDARY OUTCOMES:
cost-effectiveness ratio (ICER) between the two technologies and the 95% confidence interval for the ICER | 6 months, 1 year, 2 years
percentage of patients whose Coumadin is stopped prematurely due to inappropriate assumption of rhythm control | 6 months, 1 year, 2 years
percentage of patients who develop symptoms of stroke or transient ischemic attacks during follow up | 6 months, 1 year, 2 years
cost differences in follow up care between the two groups | 6 months, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjuya Lakkireddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States